CLINICAL TRIAL: NCT04575701
Title: Long-term Outcome of TNF Alpha Therapy in IBD
Status: Completed | Type: Observational
Sponsor: Medical University of Graz (Other)
Responsible Party: Sponsor
Other Study IDs: 1465/2018
Record Dates: First submitted 2020-09-29; First posted 2020-10-05 (Actual); Last update posted 2021-02-25 (Actual); Status verified 2021-02

CONDITIONS: IBD

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Ulcerative Colitis (UC): This Group includes all patients suffering from UC who have been treated with a TNF Alpha antibody within the last 20 years at the IBD outpatient clinic at our Hospital.
  Interventions: Other: TNF Alpha therapy
- Crohn's disease (CD): This Group includes all patients suffering from CD who have been treated with a TNF Alpha antibody within the last 20 years at the IBD outpatient clinic at our Hospital.
  Interventions: Other: TNF Alpha therapy
- IBD unclassified: This Group includes all patients suffering from IBD unclassified who have been treated with a TNF Alpha antibody within the last 20 years at the IBD outpatient clinic at our Hospital.
  Interventions: Other: TNF Alpha therapy

INTERVENTIONS:
Other: TNF Alpha therapy — Retrospective analysis of outcome of first TNF Alpha therapy

SUMMARY:
The aim of this retrospective study is to assess the outcome of patients with inflammatory bowel disease (IBD) under TNF-alpha antibody therapy over a period of 20 years

DETAILED DESCRIPTION:
Long-term results published so far show that over the years a large part of patients have to stop TNF Alpha antibody therapy in IBD. Reasons are mostly loss of effectiveness or intolerance or side effects. Reasons for the termination are usually poorly characterized with regard to the exact reason and time. As a consequence, the aim of this retrospective study is to assess the outcome of patients with inflammatory bowel disease under TNF-alpha antibody therapy over a period of 20 years

ELIGIBILITY:
Inclusion Criteria:

* Patients with a confirmed IBD diagnosis
* TNF Alpha antibody therapy in the last 20 years at our outpatient clinic

Exclusion Criteria:

* Not Meeting the inclusion criteria
* Lack of clinical data, no follow up available

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study Population includes all patients with a confirmed IBD diagnosis who have been treated with an TNF Alpha antibody in the last 20 years at our outpatient clinic in Graz, Austria
Sampling Method: Non-Probability Sample
Enrollment: 538 (Actual)
Dates: Start 2019-05-01 (Actual); Primary Completion 2020-06-01 (Actual); Study Completion 2020-07-01 (Actual)

PRIMARY OUTCOMES:
Length of first TNF Alpha Therapy in IBD patients | 20 years
  The main endpoint of this retrospective Analysis is the length of Treatment with the first TNF Alpha therapy in IBD

SECONDARY OUTCOMES:
Rate of further biologicals after first TNF Alpha therapy | 20 years
  Follow-up drug therapy after termination of TNF Alpha therapy
Rate of surgical interventions after first TNF Alpha | 20 years
  Resections after the termination of first TNF Alpha therapy
Reasons for discontinuing therapy | 20 years
  Loss of response, side effects etc.
Predictive factors | 20 years
  Predictive factors for long-term response (BMI, CRP, Alb etc.)
Number of side effects | 20 years
  Side effects of the primarily used TNF-alpha antibodies leading to discontinuation of the drug

CONTACTS AND LOCATIONS:
Overall Officials: Wolfgang Petritsch, Prof, Principal Investigator — Meduni Graz
Locations (1):
- Medical University of Graz, Graz, Austria

IPD SHARING:
Plan to Share IPD: No